CLINICAL TRIAL: NCT05757336
Title: Explore the Efficacy and Safety of Sintilimab Plus Bevacizumab Combined With Gemcitabine and Albumin-paclitaxel (AG Regimen) in First-line Treatment of Initial Unresectable Gallbladder Cancer: a Phase II Clinical Study
Brief Title: Combination of Gemcitabine, Albumin-paclitaxel , Sintilimab and Bevacizumab in Unresectable Gallbladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lu Wang, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Lu Wang, MD, PhD, Head of liver surgery department, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWK-2022-08
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Gallbladder Cancer; Initially Unresectable; the First Line Treatment
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — 130-nm albumin-bound paclitaxel; sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combined treatment group (Experimental): Combination of Gemcitabine, Nab-paclitaxel, Sintilimab and Bevacizumab GC regimen: up to the results of safety run-in stage
  * Dose A: gemcitabine 1000mg/m2, paclitaxel for injection (albumin-bound) 125mg/m2 iv Q3W
  * Dose B: gemcitabine 800mg/m2, paclitaxel for injection (albumin-bound) 100mg/m2 iv Q3W
  Sintilimab: 200mg, iv, d1, q3w Bevacizumab: 7.5mg/kg, d1, q3w
  Interventions: Drug: Combination of Gemcitabine, Nab-paclitaxel, Sintilimab and Bevacizumab

INTERVENTIONS:
Drug: Combination of Gemcitabine, Nab-paclitaxel, Sintilimab and Bevacizumab — Combination of Gemcitabine, Nab-paclitaxel, Sintilimab and Bevacizumab

SUMMARY:
Study design: Prospective, single-arm, single-center phase II clinical study; Primary endpoint: Objective response rate via investigator, Safety; Secondary endpoints: disease control rate, disease-free survival, overall survival, and proportion of acceptable radical resection of primary lesions; Main characteristics of enrolled patients: Patients with initially unresectable gallbladder cancer; Interventions: Combination of Gemcitabine, Nab-paclitaxel, Sintilimab and Bevacizumab; Sample size: Using Simon's two-stage design, 15 patients in the first stage, and if more than 4pts response, enlarge the sample size to 45 patients in total; Treatment until: 1. successfully conversed to resectable disease 2. progressed disease 3. intolerable toxicity 4. patient requests withdrawal; Research process: In this study, patients who met the inclusion criteria were evaluated at the end of every 9 weeks of treatment, up to surgical treatment or disease progression; Safety evaluation: Evaluate adverse reactions according to CTCAE 5.0; Follow up: every 90 days (±7 days) until the subject died, lost follow-up or the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Before the implementation of any trial-related procedures, sign a written informed consent 2. Male or female ≥18 years old, ≤75 years old 3. Gallbladder carcinoma confirmed by histology or cytology 4. No previous systemic anti-tumor therapy (radiotherapy, chemotherapy, targeted or immunotherapy, etc.) 5. Expected survival time > 3 months 6. At least 1 measurable lesion according to RECIST1.1 criteria 7. ECOG PS score of 0-1 8. Sufficient organ function, the subject needs to meet the following laboratory indicators:

1. Absolute value of neutrophils (ANC) ≥ 1.5x109/L and platelets ≥ 90×109/L without using granulocyte colony-stimulating factor in the past 14 days;
2. Hemoglobin > 9g/dL without blood transfusion or use of erythropoietin in the past 21 days;
3. Total bilirubin ≤ 3 × upper limit of normal (ULN);
4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are ≤2.5×ULN (patients with liver metastases are allowed ALT or AST ≤5×ULN);
5. Alkaline phosphatase (AKP) ≤2.5×ULN
6. Creatinine clearance rate (calculated using the Cockcroft-Gault formula) ≥ 50 ml/min;
7. Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN;
8. Normal thyroid function, defined as thyroid-stimulating hormone (TSH ≤ 10) within the normal range; thyroid dysfunction without clinical significance after thyroid hormone supplementation can also be included.
9. Myocardial enzyme spectrum is within the normal range (such as simple laboratory abnormalities that are judged by the investigator to have no clinical significance are also allowed to enter the group); 9. For female subjects of childbearing age, they should receive a urine or serum pregnancy test within 3 days before receiving the first study drug administration (day 1 of cycle 1) and the result is negative. If the urine pregnancy test result cannot be confirmed negative, a blood pregnancy test will be ordered. Women of non-reproductive age are defined as postmenopausal for at least 1 year, or who have undergone surgical sterilization or hysterectomy 10. If there is a risk of pregnancy, all subjects (regardless of male or female) need to use contraceptive measures with an annual failure rate of less than 1% during the entire treatment period until 120 days after the last study drug administration

Exclusion Criteria:

1. Other malignant diseases outside the biliary tract diagnosed within 5 years before the first administration (excluding radically cured skin basal cell carcinoma, skin squamous cell carcinoma, and/or radically resected carcinoma in situ, radically cured thyroid papillary carcinoma can also be included after surgery);
2. Currently participating in interventional clinical research treatment, or receiving other research drugs or using research devices within 4 weeks before the first administration;
3. Active autoimmune disease requiring systemic treatment (such as the use of disease-modifying drugs, glucocorticoids or immunosuppressants) occurred before the first dose. Replacement therapies (eg, thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy. Known history of primary immunodeficiency. Only patients with autoimmune antibody positive need to confirm whether there is an autoimmune disease according to the investigator's judgment;
4. Active hemoptysis (spitting up at least 2.5ml or 1/2 teaspoon of fresh blood) within 3 months before the first study drug administration, and active gastrointestinal bleeding within 3 months before administration;
5. Imaging shows tumor invasion/infiltration of large blood vessels or bleeding tendency assessed by researchers or radiologists;
6. Received major surgical treatment within 4 weeks before the first study drug administration (except for surgery for biopsy);
7. Severe unhealed wound ulcers or fractures;
8. Current or recent (within 10 days before receiving the first dose of the study drug) use of aspirin (>325mg/day) or other non-steroidal anti-inflammatory drugs known to inhibit platelet function for 10 consecutive days;
9. Current or recent (within 10 days before receiving the first dose of study drug) treatment with full-dose oral or parenteral anticoagulant or thrombolytic agent for 10 consecutive days Note: The prophylactic use of small doses of anticoagulants is allowed: on the premise that the international normalized ratio (INR) of prothrombin time is ≤1.5, small doses of warfarin (≤1 mg/d) and low doses of heparin are allowed for prophylactic purposes (≤12,000 U/d) or low-dose aspirin (≤100mg/d);
10. Have hereditary bleeding tendency or coagulation disorder, or history of thrombosis;
11. Are receiving systemic glucocorticoid therapy (excluding nasal spray, inhalation or other routes of topical glucocorticoid) or any other form of immunosuppressive therapy within 4 weeks before the first dose of the study Note: Physiological doses of glucocorticoids are permitted (≤10 mg/day of prednisone or equivalent)
12. There is clinically uncontrollable pleural effusion/abdominal effusion (patients who do not need drainage or stop drainage for 3 days without significant increase in effusion can be enrolled)
13. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation
14. Those who are known to be allergic to active ingredients or excipients of the study drug sintilimab, bevacizumab, gemcitabine hydrochloride for injection, paclitaxel for injection (albumin-bound type)
15. Has not recovered adequately from any intervention-induced toxicity and/or complications (ie, ≤ Grade 1 or reached baseline, excluding fatigue or alopecia) prior to initiating treatment
16. Known history of human immunodeficiency virus (HIV) infection (ie HIV 1/2 antibody positive)
17. Untreated active hepatitis B (defined as HBsAg positive and detection of HBV-DNA copy number greater than the upper limit of normal value of the laboratory laboratory of the research center)

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1. If the HBV viral load before the first administration is <2.5×103 copies/ml (500 IU/ml), the subject should receive anti-HBV treatment during the entire study treatment period
2. For subjects whose anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load are less than the upper limit of normal value in the laboratory department of the research center, they do not need to receive preventive anti-HBV treatment, but they need to be closely monitored. Monitoring for viral reactivation 18. Subjects with active HCV infection (HCV antibody positive and HCV-RNA level higher than the lower limit of detection) 19. Except for those who have received live attenuated vaccines within 4 weeks before the first dose of the new crown vaccine 20. Pregnant or lactating women 21. Esophageal or gastric variceal bleeding events caused by portal hypertension in the past 6 months; known severe (G3) varices in endoscopy within 3 months before the first administration; evidence of portal hypertension (including Imaging examination revealed that the length of splenomegaly exceeds 10 cm and the platelets are less than 100×109/L), and the researchers evaluated the risk of bleeding as high 22. Any life-threatening bleeding events occurred in the past 3 months, including the need for blood transfusion therapy, surgery or local therapy, continuous drug therapy 23. Arterial and venous thromboembolic events within the past 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis or any other serious history of thromboembolism. Implantable venous port or catheter-derived thrombosis, or superficial venous thrombosis, unless the thrombus is stabilized after conventional anticoagulant therapy 24. History of gastrointestinal perforation and/or fistula, intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colon resection or extensive small bowel resection, complicated by chronic diarrhea) within the past 6 months , Crohn's disease, ulcerative colitis, or long-term chronic diarrhea; 25. Presence of any serious or uncontrolled systemic disease, such as:

1) Resting ECG has significant abnormalities in rhythm, conduction or morphology, and the symptoms are severe and uncontrollable, such as complete left bundle branch block, heart block above second degree, ventricular arrhythmia or with fast ventricular rate atrial fibrillation 2) Unstable angina, congestive heart failure, New York Heart Association (NYHA) grade ≥ 2 chronic heart failure 3) Any arterial thrombosis, embolism or ischemia occurred within 6 months before the selected treatment, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, etc.; 4) Received major surgical operations (craniotomy, thoracotomy or laparotomy) or unhealed wounds, ulcers or fractures within 4 weeks before the first administration. Received tissue biopsy or other minor surgical procedures within 7 days before the first dose, except for venipuncture for intravenous infusion 5) Unsatisfactory blood pressure control (systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg) 6) Active tuberculosis 7) Active or uncontrolled infection requiring systemic therapy 8) Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction 9) Liver disease such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis 10) Poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L) 11) Urine routine prompts urine protein ≥ ++, and confirmed 24-hour urine protein quantity > 1.0 g; 12) Patients with mental disorders who cannot cooperate with treatment 26. Medical history or disease evidence that may interfere with the test results, prevent the subject from participating in the whole study, abnormal treatment or laboratory test values, or other situations that the investigator believes are not suitable for enrollment. The investigator believes that there are other potential risks t

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-12-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 9 weeks
  objective response rate
Safety：the incidence of adverse events and serious adverse events | 3 weeks
  Incidence of adverse events and serious adverse events

SECONDARY OUTCOMES:
disease control rate | 3 weeks
  disease control rate
progress-free survival | 3 weeks
  progress-free survival
overall survival | 3 weeks
  overall survival
Proportion of acceptable radical resection of primary lesions | 3 weeks
  Proportion of acceptable radical resection of primary lesions

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China